CLINICAL TRIAL: NCT05836506
Title: Assessment of the Relative Bioavailability of Immediate Release Formulations of ABBV-903 in Healthy Volunteers
Brief Title: A Study to Assess the Relative Bioavailability of Immediate Release Formulations of ABBV-903 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-226
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteer
Keywords: ABBV-903; Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1: Sequence A (Experimental): In Period 1 on Day 1, participants will receive ABBV-903 Tablet Form 1 after fasting. In Period 2 on Day 1, participants will receive ABBV-903 Tablet Form 2 after fasting. Lastly, in Period 3 on Day 1, participants will receive ABBV-903 Tablet Form 1 after a high fat meal. Participants will be followed up for 30 days.
  Interventions: Drug: ABBV-903 Tablet Form 1; Drug: ABBV-903 Tablet Form 2
- Part 1: Sequence B (Experimental): In Period 1 on Day 1, participants will receive ABBV-903 Tablet Form 2 after fasting. In Period 2 on Day 1, participants will receive ABBV-903 Tablet Form 1 after fasting. Lastly, in Period 3 on Day 1, participants will receive ABBV-903 Tablet Form 1 after fasting. Participants will be followed up for 30 days.
  Interventions: Drug: ABBV-903 Tablet Form 1; Drug: ABBV-903 Tablet Form 2
- Part 2: Sequence A (Experimental): In Period 1 on Day 1, participants will receive ABBV-903 Tablet Form 1 after fasting. In Period 2 on Day 1, participants will receive ABBV-903 Tablet Form 2 after fasting. Lastly, in Period 3 on Day 1, participants will receive ABBV-903 Tablet Form 2 after a high fat meal. Participants will be followed up for 30 days.
  Interventions: Drug: ABBV-903 Tablet Form 1; Drug: ABBV-903 Tablet Form 2
- Part 2: Sequence B (Experimental): In Period 1 on Day 1, participants will receive ABBV-903 Tablet Form 2 after fasting. In Period 2 on Day 1, participants will receive ABBV-903 Tablet Form 1 after fasting. Lastly, in Period 3 on Day 1, participants will receive ABBV-903 Tablet Form 2 after fasting. Participants will be followed up for 30 days.
  Interventions: Drug: ABBV-903 Tablet Form 1; Drug: ABBV-903 Tablet Form 2

INTERVENTIONS:
Drug: ABBV-903 Tablet Form 1 — Oral Tablets
Drug: ABBV-903 Tablet Form 2 — Oral Tablets

SUMMARY:
The main objective of this study is to assess the relative bioavailability and pharmacokinetics of ABBV-903 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI is ≥ 18.0 to ≤ 32 kg/m2 after rounding to the tenth.
* Negative test result for SARS-CoV-2 infection at screening visit and upon initial confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), endocrine, renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of diseases aggravated or triggered by ultraviolet radiation and no history of abnormal reaction photosensitivity or photoallergy to sunlight, or artificial source of intense light, especially ultraviolet light.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Approximately 44 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment
Maximum Plasma Concentration (Cmax) of ABBV-903 | Up to approximately 14 days
  Cmax of ABBV-903
Time to Cmax (Tmax) of ABBV-903 | Up to approximately 14 days
  Tmax of ABBV-903
Terminal Phase Elimination Half-Life (t1/2) of ABBV-903 | Up to approximately 14 days
  Terminal phase elimination half-life of ABBV-903
Area Under the Concentration-Time Curve From Time 0 to Last Measurable Concentration (AUCt) of ABBV-903 | Up to approximately 14 days
  AUCt of ABBV-903
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of ABBV-903 | Up to approximately 14 days
  AUCinf of ABBV-903

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 254926, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-226